CLINICAL TRIAL: NCT01413477
Title: Nickel Desensitization Using Topical Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Jan P. Dutz, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H10-02854
Record Dates: First submitted 2011-04-13; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatitis; Nickel allergy; Desensitization therapy
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — calcipotriene; Betamethasone; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calcipotriol ointment (Active Comparator)
  Interventions: Drug: Calcipotriol, Betamethasone, Calcipotriol & Betamethasone
- Betamethasone dipropionate ointment (Active Comparator)
  Interventions: Drug: Calcipotriol, Betamethasone, Calcipotriol & Betamethasone
- Calcipotriol and betamethasone ointment (Active Comparator)
  Interventions: Drug: Calcipotriol, Betamethasone, Calcipotriol & Betamethasone
- Vaseline Petroleum Jelly (Placebo Comparator)
  Interventions: Drug: Calcipotriol, Betamethasone, Calcipotriol & Betamethasone

INTERVENTIONS:
Drug: Calcipotriol, Betamethasone, Calcipotriol & Betamethasone — All study patients will be randomized to receive one of four topical ointments (calcipotriol, betamethasone dipropionate, combination of both calcipotriol/betamethasone dipropionate, or Vaseline petroleum jelly). Each subject will receive one unlabelled 5g tube for application to be dispensed by pharmacist, Rudy Chin. We expect approximately 2g of TOTAL use (0.125g applied twice daily over a 5 cm x 5 cm area on one forearm for 7 days). Typically, topical steroids such as betamethasone dipropionate have been used for treating a number of inflammatory skin conditions, including eczema. In addition, vitamin D analogues such as calcipotriol are used to treat psoriasis. Both agents, in our study, will be used on a small area of normal skin for a short 7 day course.
  Other Names: Dovonex (calcipotriol ointment, DIN 01976133 Leo Pharma),; Dovobet (DIN 02244126, Leo Pharma); Betamethasone diproprionate (0.5% ointment USP generic)

SUMMARY:
Nickel contact dermatitis (eczema) is one of the most common allergic conditions affecting the skin. This is a study looking at potentially desensitizing nickel-allergic patients to their allergy using anti-inflammatory ointments applied to the skin (arm). Application of these ointments (ie. modified Vitamin D) has been shown to increase specific immune cells (T regulatory cells), which play a role in preventing immune activation and subsequently inflammation. The investigators propose use of topical anti-inflammatory agents (corticosteroids, modified Vitamin D, or both) may desensitize patients with nickel allergy.

DETAILED DESCRIPTION:
1. Purpose: To evaluate whether topical anti-inflammatory ointments (calcipotriol, betamethasone dipropionate, or a combination of both) can decrease sensitivity to nickel in known nickel allergic patients. Optional blood samples will be part of the protocol to measure immune responses.
2. Hypothesis: Use of these topical agents will prevent sensitization to nickel sulfate upon re-exposure.
3. Justification: Currently, no cure can yet be offered to nickel sensitive patients. Standard treatment only involves avoiding nickel-containing products. However, this is not always easily achieved depending on patient awareness and environmental exposures. Topical desensitization has not yet been explored in patients with pre-established contact allergy. This research will be placebo-controlled with Vaseline petroleum jelly to compare reactions to nickel in those treated with anti-inflammatory ointments.
4. Objectives: a) To evaluate the use of topical anti-inflammatory agents and its role in desensitizing known nickel allergic patients to nickel. b) To measure immune cell responses to nickel allergen from a blood sample taken before and after topical anti-inflammatory application.
5. Research Method: Randomized, double-blinded, placebo-controlled, proof of principle study. Subjects meeting inclusion and exclusion criteria with known nickel sensitivity will be recruited into the study. Those who consent will undergo 3 sets of nickel patch testing: At week 1 to confirm nickel allergic status, week 3 to induce tolerance by patch testing at the site of topical ointment application, and finally at week 5 to test for desensitization. (Week 2 is self-application with topical ointment; Week 4 is a rest week).
6. Statistical Analysis: a) Primary end-point: Clinical responses measured by standard patch testing scores will be documented and photographed for comparison. b) Secondary end-point: Levels of T regulatory cell responses before and after topical treatment. c) Planned sample size: 24 patients. Given that this is a proof-of-principle study, the investigators are choosing to study a small sample size to detect any differences amongst treatment arms, if any. A larger-scale, adequately-powered study would be needed to detect any statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients have had a diagnosis of nickel allergy determined by patch testing

Exclusion Criteria:

* Treatment with immunomodulating medications concurrently or in the previous one month
* Active skin disease, particularly to the site of application (forearms)
* Hypersensitivity to calcipotriol, corticosteroids, or vehicle
* Previous anaphylactic reactions to nickel allergen
* Pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in contact dermatitis response to nickel allergen at 5 weeks after topical desensitization | All study subjects will be evaluated after each patch test session (weeks 1, 3, 5). The final outcome to assess for desensitization will be evaluated at week 5.
  Erythema, induration, blistering of the skin will be noted. The standardized Likert scale (0-3+) will be used as follows:
  1. + Weak (non-vesicular) reaction: erythema, infiltration, possibly papules
  2. ++ Strong (edematous or vesicular) reaction
  3. +++ Extreme (spreading, bullous or ulcerative) reaction
     * Negative reaction

SECONDARY OUTCOMES:
Change in immune cell profile of patients 5 weeks after nickel desensitization | All consenting subjects will have baseline blood drawn at week 0 and again at week 5 to compare any differences in immune cells (ie. T cells).
  Peripheral T cells will be separated and responses will be determined by flow cytometry after nickel desensitization therapy. Approximately 50 ml of blood will be drawn from consenting subjects. Absolute cell numbers and immunophenotypes of cells will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jan P Dutz, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Contact Dermatitis Clinic, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Ghoreishi M, Bach P, Obst J, Komba M, Fleet JC, Dutz JP. Expansion of antigen-specific regulatory T cells with the topical vitamin d analog calcipotriol. J Immunol. 2009 May 15;182(10):6071-8. doi: 10.4049/jimmunol.0804064. PMID 19414758
- [Background] Landeck L, Schalock PC, Baden LA, Neumann K, Gonzalez E. Patch-testing with the standard series at the massachusetts general hospital, 1998 to 2006. Dermatitis. 2009 Mar-Apr;20(2):89-94. PMID 19426614
- [Background] Jacob SE, Moennich JN, McKean BA, Zirwas MJ, Taylor JS. Nickel allergy in the United States: a public health issue in need of a "nickel directive". J Am Acad Dermatol. 2009 Jun;60(6):1067-9. doi: 10.1016/j.jaad.2008.11.893. Epub 2009 Jan 23. No abstract available. PMID 19167779
- [Background] Thyssen JP, Linneberg A, Menne T, Johansen JD. The epidemiology of contact allergy in the general population--prevalence and main findings. Contact Dermatitis. 2007 Nov;57(5):287-99. doi: 10.1111/j.1600-0536.2007.01220.x. PMID 17937743
- [Background] Hanneman KK, Scull HM, Cooper KD, Baron ED. Effect of topical vitamin D analogue on in vivo contact sensitization. Arch Dermatol. 2006 Oct;142(10):1332-4. doi: 10.1001/archderm.142.10.1332. PMID 17043189
- [Background] Moed H, von Blomberg BM, Bruynzeel DP, Scheper RJ, Gibbs S, Rustemeyer T. Regulation of nickel-induced T-cell responsiveness by CD4+CD25+ cells in contact allergic patients and healthy individuals. Contact Dermatitis. 2005 Aug;53(2):71-4. doi: 10.1111/j.0105-1873.2005.00635.x. PMID 16033398
- [Background] Wu X, Roelofs-Haarhuis K, Zhang J, Nowak M, Layland L, Jermann E, Gleichmann E. Dose dependence of oral tolerance to nickel. Int Immunol. 2007 Aug;19(8):965-75. doi: 10.1093/intimm/dxm066. Epub 2007 Aug 13. PMID 17698564
- [Background] Cavani A, Nasorri F, Ottaviani C, Sebastiani S, De Pita O, Girolomoni G. Human CD25+ regulatory T cells maintain immune tolerance to nickel in healthy, nonallergic individuals. J Immunol. 2003 Dec 1;171(11):5760-8. doi: 10.4049/jimmunol.171.11.5760. PMID 14634084
- [Background] Kang Y, Xu L, Wang B, Chen A, Zheng G. Cutting edge: Immunosuppressant as adjuvant for tolerogenic immunization. J Immunol. 2008 Apr 15;180(8):5172-6. doi: 10.4049/jimmunol.180.8.5172. PMID 18390698
- [Background] Zaunders JJ, Munier ML, Seddiki N, Pett S, Ip S, Bailey M, Xu Y, Brown K, Dyer WB, Kim M, de Rose R, Kent SJ, Jiang L, Breit SN, Emery S, Cunningham AL, Cooper DA, Kelleher AD. High levels of human antigen-specific CD4+ T cells in peripheral blood revealed by stimulated coexpression of CD25 and CD134 (OX40). J Immunol. 2009 Aug 15;183(4):2827-36. doi: 10.4049/jimmunol.0803548. Epub 2009 Jul 27. PMID 19635903